CLINICAL TRIAL: NCT02758353
Title: Scaling up the Use of Sulphadoxine-Pyrimethamine for the Preventive Treatment of Malaria in Pregnancy: Results and Lessons on Scalability, Costs and Program From Three Local Government Areas in Sokoto State, Nigeria
Brief Title: The Impact of Sulphadoxine-Pyrimethamine Use At Scale on Newborn Outcomes in Nigeria
Acronym: MIPP-NG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JSI Research & Training Institute, Inc. (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Federal Ministry of Health, Nigeria (Other Government)
Responsible Party: Principal Investigator, Nosa Orobaton, Senior Advisor, Global Health/Chief of Party, JSI Research & Training Institute, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: JSI-MIPP-NG #1
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Malaria; Stillbirths
Keywords: Malaria in Pregnancy; Nigeria; Sulfadoxine-Pyrimethamine; Scale up; Primary Health Care
MeSH Terms: conditions — Malaria; Stillbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Community distribution of SP (Experimental): All the eligible pregnant women were reached with SP either at health clinic and/or at community/household level with sulphadoxine-pyrimethamine (SP). Alerts and reminders were sent to them by community-based health volunteers ahead of subsequent SP doses.
  Interventions: Drug: Community distribution of SP

INTERVENTIONS:
Drug: Community distribution of SP — SP delivered at both the community and facility level by trained CBHVs in three LGAs.
  Other Names: Community Distribution of SP to eligible participants

SUMMARY:
The purpose of this study is to test the feasibility of the scale-up of sulphadoxine- pyrimethamine (SP) for the preventive treatment of malaria in pregnancy in three Local Government Areas (LGAs) in Sokoto State, Nigeria. The scale-up strategy tested included the introduction of community-based distribution of SP in addition to ongoing health facility distribution during antenatal care (ANC) visits. In addition, the study examined for the effect of SP use by participants during pregnancy on the head circumference of live newborns and on the odds of a baby being a stillborn. Finally, the investigators also sought to quantify the costs associated with program scale up SP to deliver at least three doses of SP per participant via a government operated distribution program.

DETAILED DESCRIPTION:
Study Objectives

The study objectives were to:

1. Examine scale-up mechanisms that enable increased SP coverage through community-based primary health care delivery, without reducing facility uptake of SP.
2. Examine community acceptance of SP and the likelihood of long-term community-sustained demand.
3. Document associations, if any, between increased SP coverage and improved intrauterine conditions for newborn, as measured by head circumference increments and declines in still birth rates.
4. Estimate the costs of delivering SP at scale per woman for a three doses or higher regimen.

Study Location and Relevant Contextual Information

The study was undertaken in four LGAs: Dange Shuni Goronyo and Silame (combined 2015 population, according to official Sokoto State estimates = 661,606) LGAs which were purposively selected as intervention LGAs; and Yabo LGA, the fourth (2015 population, according to official Sokoto State estimates = 167,971), was purposively selected as the counterfactual LGA. The selection criteria were that all LGAs had a high prevalence of malaria in pregnancy and that at one LGA each in the intervention group, was selected from each of the State's three senatorial zones.

Sampling Size Considerations

Given the intention of the study to examine the prospects of scaling up an already existing program, to reach all eligible pregnant participants, no sampling regimen was included in this study.

Data Collection Procedures

The community-based health volunteer (CBHV) system has an inbuilt data collection system managed by a community drug keeper (CDK) and a supervising facility-based health worker to monitor distribution at the community level. Investigators used an outcome form to collect data. Data captured in the outcome form included the condition of the newborn and mother at birth, of the newborn at birth-live birth or stillbirth-at days 7, 14 and 28 postpartum. For this study, the investigators modified the outcome form to also capture the number of SP doses a participant received and date/month the participant got them. The modified outcome form also collected data on a pregnant participant's primipara status, ANC status, gestation in months at time of delivery, the state of newborns (live or stillborn), sex of the newborn and head circumference measurements.

Nominal cost and expense data in 2015 Nigerian Naira (NGN) directly related to community and facility distribution of SP in the intervention and counterfactual LGAs were obtained from project records and other sources. The cost estimates obtained are what it would cost the state government and LGAs as de facto providers of primary health care in Nigeria, to deliver SP-related services at both the community and facility level, including start-up costs. Six cost centers were included in the analyses: health facility, LGA technical administration, CBHV supervisors, ward development committees, CBHV, and logistics for SP distribution.

Data Quality Procedures

Twelve teams of four data quality auditors, independent of other project staff, were recruited to track data quality obtained from communities. Each team comprised of three females and one supervisor. Over the life of the project, the teams visited all the participants recorded with at least one birth-that occurred during the project-in the 42 wards of the three intervention and one counterfactual LGAs. The data auditors also sought for and compiled information on omitted mothers and births. The auditors were expected to directly inquire of a participant-or an informed family member - in the event of a maternal death-if a CBHV and CBHV Supervisor visited, the status of newborns, alive or stillborn, and if head circumference was measured within seven days among live births. With participants' responses as the gold standard, births, status of births, and confirmed head circumference measurements were verified.

Statistical Analyses

Programmatic data was used to assess the coverage of SP doses during pregnancy in the intervention and counterfactual LGA's. Univariate and multivariate analyses were used by investigators to test associations between doses of SP and newborn head circumference and the odds of stillbirth. These analyses were conducted in Statistical Analysis System (SAS) v.9 and excel.

For cost data, the investigators calculated two ratios: cost per dose and cost per woman served, disaggregated by number of SP doses in the intervention and and counterfactual group. Analyses were conducted in Excel®.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be pregnant.
2. Pregnant participants must have experienced quickening in course of gestation.
3. Participants must reside in an intervention or a counterfactual LGA.

Exclusion Criteria:

1. Non-pregnant residents in a counterfactual or an intervention LGA.
2. Non-residents of counterfactual or intervention LGA.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31493 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants that got SP coverage among all pregnant women | Up to 7 months
  The percentage SP coverage among all pregnant participants and by number of SP doses ingested. The outcome form will be used to obtain an aggregate number of women that received SP. The total number of eligible women will be obtained from either an enumeration of eligible women in the intervention LGA, or by population estimation in the counterfactual LGA.

SECONDARY OUTCOMES:
Cost per Woman served with SP in Nigeria Naira | Up to 7 months
  This will be obtained from costing data produced by the study and the total number of participants served as derived from the outcome forms.
Cost per SP dose delivered in Nigeria Naira | Up to 12 months
  This will be obtained from costing data produced by the study and the total number of SP doses given as derived from the outcome forms.
Incidence of Stillbirths in stillbirths per 1000 term births | Up to 7 months
  Stillbirth is a delivery that occurred after 7 months of gestation in which a baby was birthed without any signs of life (no breathing, no movement, and no sound) as reported by a participant or an informed family member.
Head circumference of Newborn in millimeters | Up to 7 months
  Head circumference of live newborns was measured within 7 days postpartum by CBHV. The information will be aggregated from individual outcome forms.

CONTACTS AND LOCATIONS:
Overall Officials: Nosa G Orobaton, MD, DrPH, Principal Investigator — John Snow, Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] WHO. World Malaria Report 2015 [Internet]. 2015. Available from: http://apps.who.int/iris/bitstream/10665/200018/1/9789241565158_eng.pdf?ua=1
- [Background] Dellicour S, Tatem AJ, Guerra CA, Snow RW, ter Kuile FO. Quantifying the number of pregnancies at risk of malaria in 2007: a demographic study. PLoS Med. 2010 Jan 26;7(1):e1000221. doi: 10.1371/journal.pmed.1000221. PMID 20126256
- [Background] Partnership RBM. Roll Back Malaria Annual Report 2013 [Internet]. [cited 2016 Feb 21]. Available from: http://www.rollbackmalaria.org/files/files/resources/RBM-Annual-Report- 2013(1).pdf
- [Background] Onwujekwe O, Chima R, Okonkwo P. Economic burden of malaria illness on households versus that of all other illness episodes: a study in five malaria holo-endemic Nigerian communities. Health Policy. 2000 Nov 17;54(2):143-59. doi: 10.1016/s0168-8510(00)00105-6. PMID 11094267
- [Background] Desai M, ter Kuile FO, Nosten F, McGready R, Asamoa K, Brabin B, Newman RD. Epidemiology and burden of malaria in pregnancy. Lancet Infect Dis. 2007 Feb;7(2):93-104. doi: 10.1016/S1473-3099(07)70021-X. PMID 17251080
- [Background] Radeva-Petrova D, Kayentao K, ter Kuile FO, Sinclair D, Garner P. Drugs for preventing malaria in pregnant women in endemic areas: any drug regimen versus placebo or no treatment. Cochrane Database Syst Rev. 2014 Oct 10;2014(10):CD000169. doi: 10.1002/14651858.CD000169.pub3. PMID 25300703
- [Background] Blencowe H, Cousens S, Jassir FB, Say L, Chou D, Mathers C, Hogan D, Shiekh S, Qureshi ZU, You D, Lawn JE; Lancet Stillbirth Epidemiology Investigator Group. National, regional, and worldwide estimates of stillbirth rates in 2015, with trends from 2000: a systematic analysis. Lancet Glob Health. 2016 Feb;4(2):e98-e108. doi: 10.1016/S2214-109X(15)00275-2. Epub 2016 Jan 19. PMID 26795602
- [Background] Villar J, Cheikh Ismail L, Victora CG, Ohuma EO, Bertino E, Altman DG, Lambert A, Papageorghiou AT, Carvalho M, Jaffer YA, Gravett MG, Purwar M, Frederick IO, Noble AJ, Pang R, Barros FC, Chumlea C, Bhutta ZA, Kennedy SH; International Fetal and Newborn Growth Consortium for the 21st Century (INTERGROWTH-21st). International standards for newborn weight, length, and head circumference by gestational age and sex: the Newborn Cross-Sectional Study of the INTERGROWTH-21st Project. Lancet. 2014 Sep 6;384(9946):857-68. doi: 10.1016/S0140-6736(14)60932-6. PMID 25209487
- [Background] Menendez C, Ordi J, Ismail MR, Ventura PJ, Aponte JJ, Kahigwa E, Font F, Alonso PL. The impact of placental malaria on gestational age and birth weight. J Infect Dis. 2000 May;181(5):1740-5. doi: 10.1086/315449. Epub 2000 May 15. PMID 10823776
- [Background] McClure EM, Goldenberg RL, Dent AE, Meshnick SR. A systematic review of the impact of malaria prevention in pregnancy on low birth weight and maternal anemia. Int J Gynaecol Obstet. 2013 May;121(2):103-9. doi: 10.1016/j.ijgo.2012.12.014. Epub 2013 Mar 13. PMID 23490427
- [Background] WHO. Consensus Statement: Optimizing the Delivery of Malaria-inPregnancy Interventions [Internet]. 2013 [cited 2016 Feb 21]. Available from: http://www.pmi.gov/docs/default-source/default-document-library/toolscurricula/consensusreport_malariapregnancy.pdf?sfvrsn=4
- [Derived] Orobaton N, Austin AM, Abegunde D, Ibrahim M, Mohammed Z, Abdul-Azeez J, Ganiyu H, Nanbol Z, Fapohunda B, Beal K. Scaling-up the use of sulfadoxine-pyrimethamine for the preventive treatment of malaria in pregnancy: results and lessons on scalability, costs and programme impact from three local government areas in Sokoto State, Nigeria. Malar J. 2016 Nov 4;15(1):533. doi: 10.1186/s12936-016-1578-x. PMID 27814763